CLINICAL TRIAL: NCT02239042
Title: Effect of Gallium-Aluminum-Arsenide Laser - AsGaAl Low-level Laser Therapy on the Healing of Human Palate Mucosa After Connective Tissue Graft Harvesting: Randomized Clinical Trial
Brief Title: Effect of Low-level Laser Therapy on Palatal Wound Healing
Acronym: LLLT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Researcher - Principal investigator, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132.831
Record Dates: First submitted 2014-09-02; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Palatal Wound
Keywords: Gingival recessions
MeSH Terms: conditions — Gingival Recession | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-level laser therapy (LLLT) Sham (Sham Comparator): LLLT Sham on the palatal donor site of connective tissue graft
  Interventions: Procedure: LLLT
- Low-level laser therapy (LLLT) (Experimental): LLLT on the palatal donor site of connective tissue graft
  Interventions: Procedure: LLLT

INTERVENTIONS:
Procedure: LLLT — The patients allocated for the test group received the following protocol for laser application: Five (5) points of irradiation were performed. The irradiation was performed with a ASGaAl diode laser that continuously emitted a wavelength of 660 nm. 30 mW was used for 20 seconds, and the total applied energy density (fluence) was 15 J/cm2 (3 J/cm2 per point and an application time of 4 seconds per point). The applications were performed using punctual contact (to reduce reflection) with the tip perpendicular to the gingival tissue. Laser therapy was initiated in the immediate postoperative period (just after sutures) and was followed by seven more applications performed every other day, with a total of 8 laser applications. The power of the equipment was calibrated prior to each application. The patients allocated to the control group received sham irradiation. For this, black rubber protection was placed at the tip of the laser device, which did not allow the light to reach the tissue
  Other Names: Low-level laser therapy (LLLT) after Coronally advanced falp and connective tissue graft technique to treat gingival recessions on the donor site

SUMMARY:
The aim of the present study was to evaluate the influence of LLLT on the recovery of the palatine donor site wounds after harvest connective tissue graft.

DETAILED DESCRIPTION:
This was a prospective, parallel and controlled clinical trial. The population evaluated in this study was selected at Science and Technology Institute - ICT - São José dos Campos, College of Dentistry

The selected patients were randomly allocated (by a computer generated list) into:

* Group 1 (Test, n=16): Periodontal surgery for root coverage through connective tissue graft and LLLT on donor site.
* Group 2 (Control, n=16): Periodontal surgery for root coverage through connective tissue graft and LLLT SHAM on donor site.

Surgical procedure was performed by one surgeon. The gingival recession defects were treated by connective tissue graft technique. A connective tissue graft was removed from palate mucosa following Bruno technique. Briefly, a first incision on the palate was performed perpendicularly to the long axis of the teeth, 2 to 3 mm apical to the gingival margin. The mesiodistal length of the incision was determined by the length of the graft required to cover the recession. Since the selected recessions were in maxillary canines and premolars, the length of the graft vary minimally (10-12mm). The second incision was made parallel to the first one, 1-2mm apically, and parallel to the long axis of the teeth in order to separate the subepithelium connective tissue from the epithelial layer. The incision is carried far enough apically to provide a 7mm height of connective tissue to cover the denuded root surface. Afterwards, another incision parallel to the long axis of the teeth, starting from the first incision was performed to separate the subepithelium connective tissue from the periosteum. Then, the connective tissue graft was removed from the palate as atraumatically as possible. Single sutures were made on the palate (4-0 silk) and the graft was sutured on the receptor site

Clinical parameters were assessed at baseline and 7, 14, 45, 60 and 90 days post-operatively

Statistical Analysis The null hypothesis considered in the study was the absence of difference in the clinical parameters between the different groups. For data analysis, the statistical program was used. The demographic and clinical data were compared between the groups using Student's t-test. The data were first analyzed for homogeneity using the Shapiro-Wilk test, which indicated non-normal distribution. . Those presenting Shapiro-Wilk p values < 0.05 were analyzed using a Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). For remaining wound area, tissue colorimetry, tissue thickness, and post-operative discomfort parameter analysis, Two Way Repeated Measures ANOVA was performed for intra and intergroup analysis. T-test was used for intergroup comparison of number of analgesics taken. Presence or absence of scar was measured by Q-square test. For all tests significance level of 5% was used.

ELIGIBILITY:
Inclusion Criteria:

* Patients that were 20 to 70 years old, both genders; presenting gingival recession Class I or II Miller, on vital canines or pre-molars, palatine region (donor site) with no pathological or morphological alterations; patients who agreed with and signed the formal consent to participate in the study, after receiving an explanation of risks and benefits, by an individual who was not a member of the present study (Resolution no. 196 - October, 1996, and Ethics and Code of Professional Conduct in Dentistry - CFO 179/93).

Exclusion Criteria:

* Patients with systemic problems that contraindicated surgical procedure; patients under medication that would interfere with the wound healing; patients who smoked; patients who were pregnant or lactating; patients who had had periodontal surgery on the study area.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in the Remaining wound area (RWA) | 7, 14, 45 and 60 post-operative days
  For this, standardized photographs were taken (brightness, distance and angle). A scale was used as a reference to measure this area. Theses photographs were exported to image software (Image J - NIH, Bethesda, USA) and the wound area was measured in square millimeters

SECONDARY OUTCOMES:
Post-operative discomfort | 7, 14, 45 and 60 days after surgical procedure
  After air spray application, patients were required to fill a visual analogue scale (VAS), of 100mm, where the scale extremes were "no pain" to "extreme" to report measurement discomfort.

OTHER OUTCOMES:
Tissue thickness | Before and 90 days after surgery
  Through four fixed points (5mm and 7mm distant to gingival margin) from the operated region, tissue thickness of palatine masticatory mucosa before the procedure and 3 months after the procedure were assessed. One stent was made to standardize the points to be measured. The stent was positioned and, with a periodontal probe, the points were marked. Then the stent was removed and measures were made. For this, an endodontic spacer with a rubber cursor was put on the marked points for it to reach palatine bone plate. Then the cursor was taken to the tissue, not pressuring it. The distance between the spacer tip to the cursor was measured using a digital caliper

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Santamaria, DDS, Ms, PhD, Principal Investigator — FOSJC-UNESP
Locations (1):
- Fosjc-Unesp, São Jose Dos Campos/ SP, Non-US Resident, Brazil

REFERENCES:
- [Derived] Dias SB, Fonseca MV, Dos Santos NC, Mathias IF, Martinho FC, Junior MS, Jardini MA, Santamaria MP. Effect of GaAIAs low-level laser therapy on the healing of human palate mucosa after connective tissue graft harvesting: randomized clinical trial. Lasers Med Sci. 2015 Aug;30(6):1695-702. doi: 10.1007/s10103-014-1685-2. Epub 2014 Nov 6. PMID 25373688